CLINICAL TRIAL: NCT04404972
Title: Incidence of Complications in Brain Death Organ Donors. Retrospective Observational Study.
Brief Title: Incidence of Complications of Brain Death
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ondrej Hrdy, Principal Investigator, Brno University Hospital
Other Study IDs: CT0012020
Record Dates: First submitted 2020-05-22; First posted 2020-05-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Brain Death
Keywords: Brain Death; Organ Donation
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to describe the incidence of complications in brain death adult organ donors.

DETAILED DESCRIPTION:
Pathophysiological changes following brain death may complicate the care of brain death donors. These complications negatively affects function of donated organs. Understanding these complications and its incidence is crucial for their appropriate management. The aim of this retrospective observational study is to evaluate the incidence of complications in adult brain death organ donors. Date will be collected from medical records of eligible patients admitted to intensive care unit for suspected brain death in whom brain death was confirmed and who become organ donors.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* confirmed brain death
* organ donor

Exclusion Criteria:

- age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patinets with confirmed brain death admitted to university hospital who become brain death organ donor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Hypotension | 48hours prior confirmation of brain death to ICU discharge
  Hypotension is defined as increase of vasoactive drug dose by 20% or systolic blood pressure lower than 90 mmHg or need for fluid resuscitation after initial normovolemia was achieved
Serum lactate level | 48hours prior confirmation of brain death to ICU discharge
  Maximal lactate level will be evaluated during ICU stay
Catecholamine storm | 48hours prior confirmation of brain death to ICU discharge
  Catecholamine storm is defined as onset of tachycardia and/or hypertension
Myocardial dysfunction | 48hours prior confirmation of brain death to ICU discharge
  Myocardial dysfunction is defined as left ventricle ejection fraction under 50% on trans-thoracic echocardiography or S-T segment depression or elevation or T wave negativity or positive troponin serum level
ARDS | 48hours prior confirmation of brain death to ICU discharge
  ARDS is defined and stratified according to Berlin definition
Oxygenation index | 48hours prior confirmation of brain death to ICU discharge
  Oxygenation index will be calculated as PaO2 divided by FiO2
Diabetes insipidus | 48hours prior confirmation of brain death to ICU discharge
  Diabetes insipidus is defines as urine output more than 4ml/kg per hour or urine specific gravity under 1010
Renal dysfunction | 48hours prior confirmation of brain death to ICU discharge
  Renal dysfunction is defined as presence of at least one of these criteria: absolute increase in serum creatinine ≥0.3 mg/dL (≥26.4 μmol/L) or increase in serum creatinine ≥1.5x above baseline or oliguria (urine output <0.5 mL/kg per hour) for >6 hours
Coagulopathy | 48hours prior confirmation of brain death to ICU discharge
  Coagulopathy is defined as international normalised ratio above 1,5 or platelet count below 100 000 per microliter
Hypothermia | 48hours prior confirmation of brain death to ICU discharge
  Body temperature below 36°C or need for external warming

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, MD, PhD, Study Chair — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No